CLINICAL TRIAL: NCT05080478
Title: Effects of P2Y12 Receptor Inhibitors on Central and Peripheral Chemoreceptors' Sensitivity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Principal Investigator, Stanisław Tubek, Medical Doctor, Wroclaw Medical University
Other Study IDs: PREL.E190.18.004
Record Dates: First submitted 2021-09-28; First posted 2021-10-15 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Dyspnea
MeSH Terms: conditions — Dyspnea | interventions — Clopidogrel; Ticagrelor

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: patients receiving ticagrelor 90mg bid
  Interventions: Drug: Clopidogrel, Ticagrelor
- Group B: patients receiving clopidogrel 75mg qd
  Interventions: Drug: Clopidogrel, Ticagrelor

INTERVENTIONS:
Drug: Clopidogrel, Ticagrelor — P2Y12 inhibitors are prescribed following the PCI procedure in patients. Patients are enrolled on the study before administration of the first dose of the drug. Parameters are measured before and after drug initiation.

SUMMARY:
Research project objectives: Most common complication of P2Y12 inhibitors treatment, particularly with ticagrelor, is dyspnea reported in 0 to 9.3% and in 10 to 38.6% of patients taking clopidogrel and ticagrelor respectively. Pathogenesis of the P2Y12 inhibitors-induced dyspnea is unknown; however, recently published case reports suggests activation of chemosensory areas. The primary objective of this study is to assess the influence of most commonly used in clinical practice P2Y12 inhibitors - ticagrelor and clopidogrel - on central and peripheral chemosensitivities. The secondary objective of the study is to define the relationship between baseline chemosensitivity (assessed before the drug initiation) and the occurrence of dyspnea after the drug administration.

Methodology: Patients undergoing percutaneous coronary angioplasty (PCI), who according to current European Cardiac Society Guidelines are prescribed with various P2Y12 inhibitors (drug choice depends on individual clinical situation), will be enrolled to the study. Patients will be assigned to 2 groups depending on the type of P2Y12 inhibitor prescribed: Group A -patients receiving ticagrelor, Group B -patients receiving clopidogrel. In both groups chemosensitivity assessment will be performed before P2Y12 inhibitor administration and after the drug initiation. Patients will be additionally asked to fill the questionnaire regarding dyspnea sensation during the treatment (VAS scale and investigator-designed questionnaire). Peripheral chemosensitivity assessment will be performed using transient hypoxia method, when progressive hypercapnic test will be employed to test central chemosensitivity. Blinded recordings of chemosensitivity tests will be analyzed by researcher not involved in data collection. Chemosensitivities prior to and after drugs initiation will be compared separately for groups A and B using appropriate statistical tests. The results of dyspnea sensation questionnaire will be compared between patients with high- and low- peripheral chemosensitivity (assessed before P2Y12 inhibitor initiation) within particular groups.

ELIGIBILITY:
Inclusion Criteria:

* Stable coronary artery disease scheduled for invasive treatment
* Age 18 - 80 years
* Planned treatment with ticagrelor or clopidogrel (according to European Cardiology Society guidelines)

Exclusion Criteria:

* Hypersensitivity to ticagrelor or clopidogrel
* Active pathological bleeding
* History of intracranial haemorrhage
* Severe hepatic impairment
* Other contraindications to the use of ticagrelor or clopidogrel
* A need for oral anticoagulation therapy
* Concomitant therapy with a strong cytochrome P-450 3A inhibitor or inducer
* Untreated, clinically significant bradycardia or atrio-ventricular conduction disorders
* Patients requiring haemodialysis
* Clinically significant anemia and/or thrombocytopenia
* Pregnancy or breastfeeding
* Scheduled coronary artery bypass grafting (CABG)
* Any severe valvular heart disease requiring further interventional or surgical treatment
* Symptomatic bronchial asthma
* Chronic obstructive pulmonary disease (COPD) in stage C or D according to GOLD
* Carotid artery stenting, carotid endarterectomy in medical history
* NYHA IV heart failure patients
* Any mental disorder, that may influence on patient's compliance
* Any other, unmentioned here factor, which in the opinion of investigator may increase the risk of the procedures performed during the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized due to stable coronary artery disease and scheduled for interventional treatment in Hear Diseases Clinic of Wroclaw Medical University will be invited to enter the study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
The influence of P2Y12 inhibitors on peripheral and central chemosensitivity | up to 5 weeks
  Absolute change in central and peripheral chemosensitivities separately for groups A and B

CONTACTS AND LOCATIONS:
Locations (1):
- Wroclaw Medical University, Wroclaw, Lower Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided